CLINICAL TRIAL: NCT03477032
Title: Faecal Transplantation in Inflammatory Bowel Disease
Brief Title: FMT in Inflammatory Bowel Disease
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: St Vincent's Hospital Melbourne (Other)
Responsible Party: Principal Investigator, Michael Kamm, Professor, St Vincent's Hospital Melbourne
Other Study IDs: St Vincent's Hospital
Record Dates: First submitted 2018-03-19; First posted 2018-03-26 (Actual); Last update posted 2019-05-29 (Actual); Status verified 2019-05

CONDITIONS: Faecal Microbiota Transplantation; Crohn Disease; Ulcerative Colitis; Microscopic Colitis
MeSH Terms: conditions — Crohn Disease; Colitis, Ulcerative; Colitis, Microscopic | interventions — Fecal Microbiota Transplantation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Biological: Faecal Microbiota Transplantation — Faeces acquired from a healthy donor
  Other Names: FMT

SUMMARY:
This is a prospective observational cohort study, over 52 weeks, evaluating the the use of faecal microbiota transplantation amongst patients with Inflammatory Bowel Disease and Microscopic Colitis

ELIGIBILITY:
Inclusion Criteria:

* Patients with inflammatory bowel disease (Crohn's disease or Ulcerative colitis) or Microscopic Colitis proven on the basis of radiology, endoscopy or histology.
* Patients with clinically and endoscopically active, Crohn's Disease, Ulcerative Colitis or Microscopic Colitis
* Patient must have attempted reasonable medical therapies to control their disease without sufficient response.
* All patients have to be capable of attending appointments, as well completing surveys and diagnostic tests for the duration of study follow up
* The patient must be able to identify a likely stool donor

Exclusion Criteria:

* Patients with an enteropathy or colitis which cannot definitively be diagnosed as Ulcerative Colitis, Crohn's disease or Microscopic colitis
* Patients with concurrent Clostridium difficile infection
* Women who are pregnant or intending to become pregnant in the near future (less than 6 months).
* Neutrophils less than 1.0 x 109/L
* Albumin less than 20g/L
* Active gastrointestinal infection as identified by testing
* A patient on steroids (prednisolone, budesonide) at a dose that cannot be safely tapered to zero within 6 weeks of initial FMT, due to the risk of adrenal insufficiency
* Short gut syndrome and/or small intestine less than 1.5m in length as measured intra-operatively
* Perforation or active internal fistulising disease or enterocutaneous fistulae.
* Any patient that the clinicians feel is incapable of participating in the safe use of FMT.
* Current use of antibiotics for any condition

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with active inflammatory bowel disease or microscopic collitis
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2018-06-01 (Actual); Primary Completion 2019-12-31 (Estimated); Study Completion 2019-12-31 (Estimated)

PRIMARY OUTCOMES:
Clinical remission as defined by Crohn's disease activity index less than 150 | 8 weeks
  CDAI <150
Clinical remission in Ulcerative colitis: Total MAYO score </= 2 | 8 weeks
  Total Mayo score of </=2, with all mayo sub-scores being 1 or less
Clinical remission in Microscopic colitis | 8 weeks
  Mean of <3 stools/day, including a mean of <1 watery stool/day over 1 week and if steroid dependent, the ability to cease steroids without increasing symptoms over baseline disease activity assessment.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Kamm, MBBS, Principal Investigator — St Vincent's Hospital Melbourne; Emily Wright, MBBS, Principal Investigator — St Vincent's Hospital Melbourne; Chamara Basnayake, MBBS, Principal Investigator — St Vincent's Hospital Melbourne; Amy Hamilton, PhD, Principal Investigator — St Vincent's Hospital Melbourne
Locations (1):
- St Vincent's Hospital, Melbourne, Victoria, Australia

IPD SHARING:
Plan to Share IPD: No